CLINICAL TRIAL: NCT06750133
Title: A Study of Universal CNK-UT Cell Injection in Patients With Refractory Acute Graft-versus-host Disease
Brief Title: Universal CNK-UT Therapy for Refractory aGVHD
Acronym: CNK-UT
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: ST Phi Therapeutics Co., Ltd (Unknown)
Responsible Party: Principal Investigator, Yi Luo, Professor, First Affiliated Hospital of Zhejiang University
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CNK-UT-IIT202305
Record Dates: First submitted 2024-12-20; First posted 2024-12-27 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Acute Graft-versus-Host Disease
Keywords: CNK-UT cell; aGVHD; allo-HSCT; steroids refractory; cellular therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CNK-UT cell Therapy (Experimental): 1. Dose Escalation：Single-dose intravenous injection of CNK-UT cells (3×10^7 CNK+ cells/kg).
  2. Dose Expansion：Multiple-dose intravenous injection of CNK-UT cells (6-10×10^7 CNK+ cells/kg)according to the results of dose escalation.
  Interventions: Biological: Chimeric Natural Killer Receptor Universal T-cells (CNK-UT)

INTERVENTIONS:
Biological: Chimeric Natural Killer Receptor Universal T-cells (CNK-UT) — Dose Escalation (Single Ascending Dose Study, SAD): During SAD study stage, the participants will be intravenous infused with CNK-UT cells (3×10^7 CNK+ cells/kg)with a"3 +3" design to determine the maximum tolerated dose. During single ascending dose (SAD) study stage, the participants will receive a single dose of CNK-UT cells before the DLT observation period (21 days). If the participants do not experience DLT, they will be able to enter a multiple ascending dose (MAD) study stage.
  Dose Expansion (multiple ascending dose study, MAD): During MAD study stage, the participants will receive multiple doses of CNK-UT cells(6-10×10^7 CNK+ cells/kg). The dosage and frequency of drug administration in the dose expansion stage can be adjusted and determined according to the SAD study.

SUMMARY:
This is a single arm, open-label, multi-center, pilot studies (Investigator Initiated Trial, IIT) to evaluate the safety, tolerability, efficacy, pharmacokinetics and pharmacodynamics of universal T-cells engineered with chimeric natural killer receptor (CNK-UT) to treat the patients with steroid-refractory/resistant or steroid-dependent aGVHD.

DETAILED DESCRIPTION:
This is a single arm, open-label, multi-center, pilot studies (Investigator Initiated Trial, IIT) to evaluate the safety, tolerability, efficacy, pharmacokinetics and pharmacodynamics of universal T-cells engineered with chimeric natural killer receptor (CNK-UT) to treat the patients with steroid-refractory/resistant or steroid-dependent acute graft-versus-host disease (aGvHD) after allogeneic hematopoietic stem cell transplantation (allo-HSCT).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 14-70 years, male or female;
2. Participants diagnosed with grade II~IV steroid-refractory/resistant or steroid-dependent aGVHD after allogeneic hematopoietic stem cell transplantation.
3. ECOG physical status score 0~3;
4. Estimated life expectancy > 12 weeks;
5. Female participants of childbearing age must undergo a serum or urine pregnancy test before enrollment, and the results must be negative, and agree to take acceptable measures to minimize the possibility of pregnancy during the trial; For female participants of childbearing age or male participants whose sexual partners are women of childbearing age, effective contraceptive measures should be taken during the study and for at least 6 months following the last dose of the study cells infusion.
6. Participants voluntarily participate in clinical trial; Understand and know this study, sign an informed consent form, and be willing to follow all experimental procedures.

Exclusion Criteria:

1. Suffering from malignant tumors or diagnosed within 5 years before enrollment, excluding radical skin basal cell carcinoma, skin squamous cell carcinoma, thyroid cancer, breast cancer (ductal carcinoma in situ) and / or radical resection of carcinoma in situ.
2. Participants with a history of organ transplantation;
3. Participants who have previously undergone more than one allogeneic hematopoietic stem cell transplantation.
4. Uncontrolled hypertension as determined by principal investigator, a history of hypertensive crisis or hypertensive encephalopathy; symptomatic congestive heart failure (New York Heart Association classification III-IV); symptomatic or poorly controlled arrhythmias; a history of congenital long QT syndrome or a corrected QT interval (QTc) > 500 ms at screening (calculated using the Fridericia method)..
5. Systemic diseases deemed unstable by principal investigator include, but are not limited to, severe pulmonary, hepatic, renal, or metabolic disorders that require pharmacological intervention (excluding complications related to allogeneic hematopoietic stem cell transplantation).
6. Active pulmonary tuberculosis (TB), who is receiving anti-tuberculosis treatment or has received anti-tuberculosis treatment within 1 year before enrollment; human immunodeficiency virus (HIV) infection, known syphilis infection.
7. Severe infections that are active or poorly controlled clinically.
8. Participants who have received treatment from other clinical trials within 12 weeks prior to the initiation of the study.
9. Participants who have previously used any gene therapy products prior to the initiation of the study.
10. Allergic to components of CNK-UT injection.
11. Participants suffer from known mental or substance abuse disorders, which may interfere with their ability to comply with research requirements.
12. Women who are pregnant or breastfeeding, as well as male or female participants who have planned for birth within 1 year after receiving medication.
13. Uncontrolled/uncorrectable metabolic disorders or other non-malignant organ diseases or systemic diseases or secondary reactions to cancer, which can lead to higher medical risk and/or uncertainty in survival assessments.
14. Other situations that the participant is identified by the investigator as unsuitable to participate in the study.

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 23 (Estimated)
Dates: Start 2024-12-14 (Actual); Primary Completion 2025-12-14 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | up to 1 year
  Incidence of Treatment Related AEs, AEs of special interest and serious adverse events (SAEs) assessed by NCI-CTCAE v5.0 criteria
Identification of Maximum Tolerated Dose (MTD) & incidence of Dose-limiting Toxicities (DLTs) | up to 21 days since first infusion of CNK-UT cells
  Incidence of dose-limiting toxicities (DLTs)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Overall response is defined as either a complete or partial response (CR+PR), the response should be confirmed no less than 4 weeks after the first evaluation.
  Overall response is defined as either a complete or partial response (CR+PR), the response should be confirmed no less than 4 weeks after the first evaluation.
Best Overall Response (BOR) | 6 months
  The best efficacy recorded from the beginning of treatment to the progression or recurrence of the disease.
Duration of Response (DOR) | 6 months
  The period from the first evaluation of CR or PR to the first evaluation of PD or death of any cause.
Progression-free Survival (PFS) | 6 months
  The period from the day when the participant receives the cell therapy to the first recorded disease progression (whether treated or not) or death of any cause, which occurs first.
Overall survival (OS) | 6 months
  The period from the first infusion to any cause of death.
Pharmacokinetics (PK) (Cmax) | up to 48 weeks
  The Peak Plasma concentration (Cmax) of amplified CNK-UT DNA in peripheral blood after infusion.
Pharmacokinetics (PK) (Tmax) | up to 48 weeks
  The time to reach the maximum concentration (Tmax)
Pharmacokinetics (PK) | up to 48 weeks
  The Area under the plasma concentration versus time curve (AUC) of amplified CNK-UT DNA in peripheral blood after infusion.
Levels of peripheral blood lymphocyte subsets | up to 48 weeks
  Percentage of CD45+CD3+TCR+T cell、CD3+CD8+ CD25+ CD69+T cell、CD3+CD4+CD25+ CD69+ T cell and Treg（CD4+CD25+FoxP3+）cell in peripheral blood detected by FCM after infusion.

OTHER OUTCOMES:
Biomarkers | Enrollment and evaluated as complete remission (CR), or if necessary，up to 48 weeks
  ST2、REG3α and Elafin will be analyzed
HLA typing | Enrollment.
  Evaluate the impact of HLA typing matching between donors and participants on the survival time and efficacy of CNK-UT in vivo.
Incidence of virus infection | up to 48 weeks
  In this study, all subjects were tested for aGVHD-associated virus infection, including cytomegalovirus and Epstein-Barr virus.
long-term survival | 5 years
  long-term survival of patients accepted universal CNK-UT cell injection therapy
Incidence of secondary tumor | 5 years
  long-term investigation of secondary tumor in patients accepted universal CNK-UT cell injection therapy

CONTACTS AND LOCATIONS:
Overall Officials: He Huang, PHD, Principal Investigator — First Affiliated Hospital of Zhejiang University
Locations (2):
- China (2):
  - First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - The first affiliated hospital of zhejiang university, school of medicine., Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes
The Clinical Study Report (CSR) and results will be shared after finish of the clinical trial.
Supporting Information: CSR
Time Frame: after the clinical trial completed
Access Criteria: contact with Principal Investigator